CLINICAL TRIAL: NCT02916303
Title: Cost-effectiveness of Early Intervention in First-episode Psychosis: Economic Evaluation of the PAFIP Program at Medium and Long-term
Brief Title: Cost-effectiveness of Interventions in First-episode Psychosis
Acronym: PAFIPEC
Status: Unknown | Type: Observational
Last Known Status: Enrolling by invitation
Sponsor: Fundación Marques de Valdecilla (Other)
Collaborators: Centro de Investigación Biomédica en Red de Salud Mental (Network); Instituto de Investigación Marqués de Valdecilla (Other)
Responsible Party: Principal Investigator, Benedicto Crespo-Facorro, Professor of Psychiatry, Fundación Marques de Valdecilla
Other Study IDs: PAFIPEC
Record Dates: First submitted 2016-07-22; First posted 2016-09-27 (Estimated); Last update posted 2020-01-14 (Actual); Status verified 2019-02

CONDITIONS: Schizophrenia
Keywords: Schizophrenia; Psychosis; Effectiveness
MeSH Terms: conditions — Schizophrenia; Psychotic Disorders

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Patients: Patients followed up at least during 3 years at PAFIP clinic

SUMMARY:
Schizophrenia has very significant economic consequences. Costs fall on many different parts of society, especially on individuals with schizophrenia and their families. The first five years after onset appears to be a critical period in which the symptoms are more responsive to treatment. In addition, if left untreated for a long time, psychosis can impact many areas of a person's life. The evidence base regarding the effectiveness of specialist early intervention services for psychosis has grown steadily and evidence from randomized controlled trials in Denmark, the United Kingdom and Spain has demonstrated the superiority of specialized early intervention programs over standard care on a broad range of outcomes including symptomatic and vocational, social functioning, and reduced inpatient care and treatment dropout, as measured over follow-up intervals of 2-3 years. Information about the cost-effectiveness of early intervention programs for first-episode psychosis is limited. The provision of such services requires investment by health departments and services, and the question of whether such services represent value for money has to date received little research attention. Only a few international studies, and none conducted in Spain, have investigated the cost effectiveness of early intervention in psychotic disorders at medium (3 years) and long-term (up to 10 years). In this study, the investigators aimed to analyse the cost-effectiveness of an intensive early-intervention programme, using data from First Episode Psychosis Clinical Program (PAFIP), the largest trial treating first episode non-affective psychosis in Spain to date.

ELIGIBILITY:
Inclusion Criteria:

* Meeting Diagnostic and Statistical Manual of Mental Disorders, Fourth Edition (DSM-IV) criteria for a principal diagnosis of schizophreniform, schizophrenia, schizoaffective, brief reactive psychosis, or psychosis non otherwise specified.
* Living in the catchment area.
* No prior treatment with antipsychotic medication or, if previously treated, a total life time of adequate antipsychotic treatment of less than 6 weeks.
* Current psychotic symptoms of moderate severity or greater assessed by one of the five items of the Scale for the Assessment of Positive Symptoms (SAPS).
* First episode patients with at least one assessement at 3 years or 10 years.

Exclusion Criteria:

* Meeting DSM-IV criteria for mental retardation.
* Meeting DSM-IV criteria for drug dependence.

Ages: 15 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Study Population: Individuals included in the First Episode Psychosis Clinical Program (PAFIP) at the University Hospital Marqués de Valdecilla (Santander - Cantabria) from February 2001.
Sampling Method: Non-Probability Sample
Enrollment: 490 (Estimated)
Dates: Start 2016-06 (Actual); Primary Completion 2017-07 (Actual); Study Completion 2020-12 (Estimated)

PRIMARY OUTCOMES:
Cost of pharmacological and non-pharmacological treatments in monetary units (€) | 3 years and 10 years

SECONDARY OUTCOMES:
Cost of inpatient treatment in monetary units (€) | 3 years and 10 years
Cost of suicide attempt in monetary units (€) | 3 years and 10 years
Burden of unemployment rate in monetary units (€) | 3 years and 10 years
Expenditure in transportation in monetary units (€) | 3 years and 10 years

CONTACTS AND LOCATIONS:
Overall Officials: Benedicto Crespo-Facorro, Professor, Principal Investigator — University Hospital Marqués de Valdecilla, IDIVAL, Department of Psychiatry, School of Medicine, University of Cantabria, Santander, Spain. CIBERSAM Centro Investigación Biomédica en Red Salud Mental, Madrid, Spain
Locations (1):
- University Hospital Marqués de Valdecilla, Santander, Cantabria, Spain

IPD SHARING:
Plan to Share IPD: No